CLINICAL TRIAL: NCT02775526
Title: Trans-Obturator Tape, Tension-Free Vaginal Tape and Burch Colposuspension for Treatment of Female Mixed Urinary Incontinence: A Randomized Clinical Trial
Brief Title: TOT, TVT And Burch Colpo-Suspension for Treatment of Female Mixed Urinary Incontinence
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Mohamed S Sweed, MD, Dr, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AS1234
Record Dates: First submitted 2016-05-15; First posted 2016-05-17 (Estimated); Last update posted 2020-01-28 (Actual); Status verified 2020-01

CONDITIONS: Treatment
Keywords: Mixed urinary incontinence; Transobturator tape (TOT); Tension-Free Vaginal Tape (TVT); Burch colposuspension; Urinary incontinence
MeSH Terms: conditions — Urinary Incontinence | interventions — Suburethral Slings

ARMS (3):
- TOT (Active Comparator): TOT
  Interventions: Procedure: TOT
- TVT (Active Comparator): TVT
  Interventions: Procedure: TVT
- Burch colposuspension (Active Comparator): Burch colposuspension
  Interventions: Procedure: Burch Colposuspension

INTERVENTIONS:
Procedure: TOT — 70 patients
  Other Names: Trans-Obturator Tape
  Arms: TOT
Procedure: TVT — 70 patients
  Other Names: Tension-Free Vaginal Tape
  Arms: TVT
Procedure: Burch Colposuspension — 70 patients
  Arms: Burch colposuspension

SUMMARY:
This prospective interventional randomized controlled trial will recruit women with MUI scheduled for surgical treatment where patients will be randomized to either Burch colposuspension, TOT or TVT. Regular postoperative follow up will be planned for at least 2 years. The primary outcome measures will be the objective and subjective cure rates.

ELIGIBILITY:
Inclusion Criteria:

* Women with mixed urinary incontinence.

Exclusion Criteria:

* Women with associated gynecological surgery e.g. uterine prolapse, previous anti-incontinence surgery, intrinsic sphincter deficiency (ISD), and medical disorders affecting the bladder innervation as diabetes mellitus were excluded from the study.
* Women who improved on medical treatment with persistence of stress element only were also excluded.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 220 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2020-01-10 (Actual); Study Completion 2020-01-10 (Actual)

PRIMARY OUTCOMES:
objective cure rate | 2 years
subjective cure rate | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Egypt